CLINICAL TRIAL: NCT07010068
Title: Nutritional Support With TGF-β2 Food for Special Medical Purposes (TGF-β2 FSMP) in Adult Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT) for the Prevention of Malnutrition: a Prospective, Randomized, Multicenter Study - (TGF-NUTRIALLO Study)
Brief Title: Nutritional Support With TGF-β2 Food for Special Medical Purposes (TGF-β2 FSMP) in Adult Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT) for the Prevention of Malnutrition: a Prospective, Randomized, Multicenter Study
Acronym: TGF-Nutri
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Enrico Morello, Enrico Morello, Principal Investigator, Head of Supportive Care Unit, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NP 6412
Record Dates: First submitted 2025-05-19; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Malnutrition (Calorie); Stem Cell Transplant Complications
Keywords: Stem Cell Transplant; malnutrution; gvhd
MeSH Terms: conditions — Malnutrition; Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, randomized, multicentric, interventional TGF-β2-enriched supplementation (Modulen IBD ®) in patients submitted to allogeneic hematopoietic stem cell transplantation (allo-HSCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MODULEN-IBD SUPPLEMENTATION (Experimental): From hospital admission to day +28 calories by Modulen-IBD® will integrate oral diet with 20% of calories by Modulen IBD® of TDEE, according to table 2 and to twice weekly monitoring
  Oral administration:
  Once reconstituted with bottled water according label instructions and at a caloric concentration of ≤1 kcal/ml, the supplement could be flavored according to the patient's tastes with barley coffee or decaffeinated coffee or cocoa. It is recommended to take in 2-3 portions to be taken throughout the day.
  NGT route:
  Placement of a small NGT (max 8-10 fr.) is recommended. Food assumption is encouraged even when NGT is placed. In case of NGT placement, the amount of calories by tube is the difference between TDEE and the amount of calories assumed with food.
  Modulen IBD® will be prepared and administered in 100-250 ml boluses (every 4-6 hours) to ensure the stability of the product.
  If a patient refuses food, Enteral Nutrition as polymeric standard, isocaloric, isoproteic, +/- fibers,
  Interventions: Dietary Supplement: TGF-β2-enriched food for special medical purposes
- BST (Best Supportive Treatment) (Active Comparator): Nutritional support in patients randomized to BST should be carried out according to EBMT-Handbook standards. If the patient's caloric intake is less than 75% for 3 days (instead 60% as proposed by EBMT manual) nutritional intervention is warranted and calculated according to BMI (see above).
  ONS: ONS should ensure the same amount of caloric intake of the experimental treatment in addition to usual food assumption. If patients could not assume the right amount of calories with ONS and refuse NGT parenteral nutrition is permitted.
  Parenteral Nutrition (PN): 3-1 formulations with a 1.1 Kal/ml content should be preferred (ex. Smofkabiven®, Olimel®) through a central line. The choice of PN type is according to the center's policy and used in combination with food or ONS assumption.
  Interventions: Dietary Supplement: BST

INTERVENTIONS:
Dietary Supplement: TGF-β2-enriched food for special medical purposes — The experimental treatment is Modulen-IBD®, a food for special medical purpose, polymeric, enriched with TGF-beta. If the patient refuses the experimental supplementation, NGT will be proposed to ensure the correct intake of Modulen-IBD® supplementation.
  If the patient refuses, not tolerates, or there are contraindications to NGT placement, best supportive therapy will be warranted as reported below (BST).
  Arms: MODULEN-IBD SUPPLEMENTATION
Dietary Supplement: BST — Best Nutritional Supportive Treatment as per center's policy according to EBMT Handbook 2024
  Arms: BST (Best Supportive Treatment)

SUMMARY:
prospective, randomized, multicenter study to confirm the potential benefits of TGF-β2 enriched FSMP. The primary objective is to evaluate the superiority of supplementing with TGF-β2 FSMP (experimental arm) compared to best supportive treatment (BST) in preventing malnutrition in patients submitted to allo-SCT. The secondary endpoints include the assessment of reduction of incidence of severe acute GVHD at day +100.

ELIGIBILITY:
Inclusion Criteria:

* Intact intestinal tract
* Life expectancy more than 12 weeks
* Allogeneic stem cell transplantation
* Signed informed consent

Exclusion Criteria:

* Active hematological disease at the beginning of conditioning
* Personal history of inflammatory bowel diseases
* Personal history of bowel resection
* Personal history of gastric bypass procedures
* Enrolment in a competitive prospective study (malnutrition or GVHD as primary outcome)
* Subjects with known hypersensitivity to milk proteins or components of Modulen-IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevention | given from day -7 to day +28
  ● PG-SGA score C (severe malnutrition) at day +28 <50%

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Morello, MD, PhD, Principal Investigator — Asst Degli Spedali Civili Di Brescia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07010068/Prot_SAP_000.pdf